CLINICAL TRIAL: NCT07015346
Title: A Non-inferiority Open-labelled Crossover Randomized Controlled Trial, of Two Arms, to Investigate the Adhesiveness and Safety of Rotigexole 8 mg/24 Hours Transdermal Patch, Manufactured by Eva Pharma, Egypt, Compared to the Innovator Product, Neupro® 8 mg/ 24 Hours Transdermal Patch, Manufactured by UCB Pharma S.A., Belgium, After 24 Hours of Application
Brief Title: Adhesion and Safety of Rotigexole Compared to Neupro®
Acronym: START
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Pharma (Industry)
Collaborators: MARC-CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: START24042025
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Rotigexole; Rotigotine; non-inferiority; open label; multicentric; randomized; cross-over
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Intervention Model Description: After signing the ICF, eligible patients will be enrolled in a 3-week run-in phase using Neupro ® gradually increasing the dose from 4 mg to 6mg then to 8 mg in weekly increments.
  Patches are applied to clean, healthy skin on rotating body sites and replaced every 24 hours, with no reuse of the same site within 14 days.
  After this phase, participants enter a 5-day intervention where they receive either Rotigexole or Neupro® in alternating sequences, with patch adhesion monitored at set intervals.
  Patients stay in a controlled setting during this phase, and patch application follows strict site rotation and documentation protocols.
  Following the intervention, patients are stabilized with Ramixole and undergo a final safety evaluation two weeks later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Rotigexole 8 mg/24 hours transdermal patch (Experimental): At the beginning of the intervention phase, patients' randomization will take place to determine the sequence of reference (R) and test (T) administration to either RTRT group or TRTR group. After obtaining all baseline characteristics, once daily patch application of one patch of 8 mg/24 h of Test (T) or Reference (R) over 4 days, i.e. a total of 4 alternating applications with RT sequence or TR sequence will be administered. Each patch remains applied for 24 h and the treatment patches may be directly switched without washout phase.
  Interventions: Drug: Rotigexole 8 mg
- Reference: Neupro® 8 mg/ 24 hours transdermal patch (Active Comparator): At the beginning of the intervention phase, patients' randomization will take place to determine the sequence of reference (R) and test (T) administration to either RTRT group or TRTR group. After obtaining all baseline characteristics, once daily patch application of one patch of 8 mg/24 h of Test (T) or Reference (R) over 4 days, i.e. a total of 4 alternating applications with RT sequence or TR sequence will be administered. Each patch remains applied for 24 h and the treatment patches may be directly switched without washout phase.
  Interventions: Drug: Neupro ® 8 mg

INTERVENTIONS:
Drug: Rotigexole 8 mg — Rotigotine 8 mg
  Other Names: Rotigotine 8 mg
  Arms: Test: Rotigexole 8 mg/24 hours transdermal patch
Drug: Neupro ® 8 mg — Rotigotine 8 mg
  Other Names: Rotigotine 8 mg
  Arms: Reference: Neupro® 8 mg/ 24 hours transdermal patch

SUMMARY:
A non-inferiority open-labelled crossover randomized controlled trial, of two arms, to investigate the adhesiveness and safety of Rotigexole 8 mg/24 hours transdermal patch, manufactured by Eva pharma, Egypt, compared to the innovator product, Neupro® 8 mg/ 24 hours transdermal patch, manufactured by UCB Pharma S.A., Belgium, after 24 hours of application

DETAILED DESCRIPTION:
Study Design: A non-inferiority open-labelled crossover randomized controlled trial, of two arms, to investigate the adhesiveness and safety of Rotigexole 8 mg/24 hours transdermal patch, manufactured by Eva pharma, Egypt, compared to the innovator product, Neupro® 8 mg/ 24 hours transdermal patch, manufactured by UCB Pharma S.A., Belgium, after 24 hours of application.

Planned Treatment Duration per Subject and Study Duration per Subject:

The overall duration of the study preparation and study conduction is 7 weeks and 5 days (54 days) that are scheduled as follows:

1. Preparatory Phase of the Study: Patients Screening (2 weeks):

   Patient screening for eligibility will occur over 14 days. During this time, all relevant administrative, demographic data collection, and informed consent will be conducted for eligible patients.
2. Run-in-Phase (3 weeks):

   * On the first day of the run-in phase, prior to drug administration, comprehensive physical and laboratory re-assessments will be conducted to document the initial patient's systemic status which will be monitored throughout the study to observe any potential systemic alterations for ethical purposes.
   * The transdermal patch Rotigotine (Neupro ®) only will be applied in the run-in phase in a dose taper manner on weekly basis according to the European Medicines Agency (1) and the US FDA (2) recommendations for treating cases of PD. A starting dose of 4 mg/24 h initially, increasing in weekly increments of 2 mg/24 h (based on clinical response and tolerability) to a maximum of 8 mg/24 h; starting dose of 4 mg/24 h in the 1st week will be applied followed by 6 mg/24 h in the 2nd week and finally 8 mg/24 h in the 3rd week.
   * The patch should be applied on clean, dry, healthy skin on the abdomen (tummy), thigh, hip, side, shoulder or upper arm.
   * A Rotigotine transdermal patch necessitates daily replacement as the drug delivery lasts for 24 hours only (3-5). Notably, re-application at the same site should be avoided for 14 days.
   * Comprehensive physical and laboratory assessments will be re-evaluated at the last day of the run-in-phase and prior to the commencement of the following intervention phase.
3. Intervention Phase of the Study:

   * This phase will last for five days only.
   * At this phase patients will be randomly assigned to sequence of TRTR or RTRT (T=Test=Rotigexole, R=Reference= Neupro ®). Each transdermal patch, either T or R, will be replaced at the same time every 24 hours.
   * Patients will receive accommodation for four nights during the intervention period to assess adhesion. Adhesion assessments will occur at 4, 8, 12 and 24 hours in accordance with FDA guidelines for transdermal patch evaluation.
   * The application of the transdermal patches should be on different sites of the same region "abdomen (tummy), thigh, hip, side, shoulder or upper arm".
   * Subjects must refrain from using topical products on the skin area designated for TDS application due to potential effects on adhesion. Additionally, hair at the application site should be clipped rather than shaved.
   * The alternating transdermal patch should then be applied on the same site of the same region on the contralateral side.
   * During this period, the patient is allowed to practice his or her routine activities without any restrictions in movement.
   * Assessments will be performed just after application and will be repeated at 4, 8, 12 and 24 hours
   * Patch reinforcement such as over-taping should be avoided.
   * At each assessment, photographic documentation of TDS adhesion to the skin must be archived. This documentation serves to corroborate the visual evaluation of adhesion percentages recorded at each time point.
   * At the final assessment of the 2nd transdermal patch application, the patient will be prescribed an alternative medicament (Ramixole) to stabilize the patient's conditions.
4. Post-intervention Phase:

   * All participants will undergo a comprehensive re-evaluation two weeks post-study to identify any systemic alterations for safety and ethical considerations (one follow-up visit).
   * Any arising adverse systemic conditions in patients will be appropriately managed

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged ≥30 years at Screening
2. Diagnosed with idiopathic Parkinson's disease with a Hoehn and Yahr stage of II to III.
3. Patients who have not received dopamine agonists in the past 30 days or are willing to discontinue current dopamine agonist therapy for the duration of the study
4. Subjects should have a Mini Mental State Examination (MMSE) score of ≥25 at Screening.
5. Participants who are able to tolerate Rotigotine transdermal patch incremental run-in period for 3 weeks.
6. Willing to refrain from swimming, bathing or sauna use on assessment days.
7. Participants should be using a reliable method of contraception (e.g., intrauterine device, barrier methods, condoms) throughout the study and for at least 30 days after the last dose of study medication
8. Female participants should have a negative pregnancy test at screening, before starting study medication and for at least 30 days after the last dose of study medication
9. Ability to provide written informed consent.

Exclusion Criteria:

1. Patients with a medical history indicating a Parkinsonian syndrome other than idiopathic PD (e.g., drug-induced, post-stroke)
2. History of significant skin hypersensitivity to adhesives or other transdermal products.
3. History of or clinical features consistent with atypical parkinsonian syndromes (e.g., multiple system atrophy, progressive supranuclear palsy)
4. CNS or psychiatric disorders other than idiopathic PD (mild depression or anxiety arising in the context of PD is not exclusionary).
5. Use of any symptomatic drug for PD other than levodopa, pramipexole, ropinirole, or Rotigotine within 60 days prior to the first dose.
6. Patients with a history of brain surgery for PD (e.g., pallidotomy, thalamotomy, deep brain stimulation).
7. Recent exposure to monoamine oxidase type A inhibitors, amphetamines, dopamine-depleting antihypertensive agents, neuroleptics, or antiemetics that block central dopamine activities.
8. Unstable or clinically significant cardiovascular disease within the last year prior to screening (e.g., arrhythmias, conduction blocks, congestive heart failure.
9. Concomitant disease or unstable medical condition within 6 months of screening that could interfere with the study or treatment.
10. Participant has history of or presence of neuroleptic malignant syndrome at screening as assessed by the investigator.
11. Participant has a current diagnosis of Epilepsy, has a history of seizures, stroke, or transient ischemic attack within 1 year prior to screening
12. Presence of hepatitis B surface antigen (HBsAg) or positive for total hepatitis B core antibody (HbcAb), or positive hepatitis C (HCV) at screening.
13. Vaccines other than SARS-CoV-2 vaccine within 28 days prior to the first dose or plans to receive vaccines during the study or within 28 days of the last dose.
14. History of immunodeficiency disease (e.g., HIV).
15. Clinically significant abnormalities in laboratory test results at screening, including hepatic and renal panels, complete blood count, chemistry panel, and urinalysis.
16. Recently unresolved allergies, hypersensitivity, contact dermatitis or an active skin disease.
17. Participants who have history of alcohol abuse within 6 months before screening as assessed by the investigator.
18. Pregnant or lactating females

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative mean percentage adhesion of the transdermal patch over the 24-hour dosing interval for two treatment periods, compared between Rotigexole (Test) and Neupro® (Reference) | two treatment periods (4 days)
  Using a mixed-effects model adjusted for period and sequence effects, with subject as a random effect

SECONDARY OUTCOMES:
Proportion of participants achieving more than 90% adherence at 4, 8, 12 and 24 hours at each period as assessed by the investigator/designee as per modified EMA scale for adhesion. | two treatment periods (4 days)
Adjusted Mean adherence percentage at each assessment time (4, 8, 12 and 24 hours). | two treatment periods (4 days)
Proportion of participants with a meaningful degree of detachment (more than half of the patch lifting off the skin or falling off) at 4, 8, 12 and 24 hours. | two treatment periods (4 days)
Number of patches that are completely detached at 4, 8, 12 and 24 hours. | two treatment periods (4 days)
Number of participants with cold flow in each treatment period (Cold flow is defined as dark ring formed around the patch). | two treatment periods (4 days)
Number of participants with patch movement/displacement in each treatment period. | two treatment periods (4 days)
Number of participants with patch wrinkling in each treatment period. | two treatment periods (4 days)
Number of participants with patch residue formation in each treatment period (Patch residue formation is assessed at patch application on the release liner and at patch removal on the skin). | two treatment periods (4 days)
% of patients reporting ease or difficulty in patch application and removal. | two treatment periods (4 days)
Frequency of Adhesion-Related Issues: Evaluate the frequency of adhesion-related issues (e.g., patch detachment). | two treatment periods (4 days)
% of patients with reported interference in daily activities due to patch adhesion. | two treatment periods (4 days)
% of patients reporting overall satisfaction with wearing each patch type, measured using a Patch Wear Satisfaction Scale. | two treatment periods (4 days)
The incidence, seriousness and severity of adverse events (AEs) including application site reactions, and discontinuations because of AEs | two treatment periods (4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem S Mohammed, Dr., Principal Investigator — Al-Manial Specialized Hospital - Cairo University; Ali S Shalash, Dr., Principal Investigator — Ain Shams Specialized Hospital - Ain Shams University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.ema.europa.eu/en/medicines/human/EPAR/neupro
- See also: Related Info — http://doi.org/10.1007/s40263-019-00646-y
- See also: Related Info — http://www.fda.gov/drugs/guidance-compliance-regulatory-information/guidances-drugs
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/31243728/8
- See also: Related Info — http://www.ema.europa.eu/contact
- See also: Related Info — http://pmc.ncbi.nlm.nih.gov/articles/PMC3900336/